CLINICAL TRIAL: NCT02105766
Title: Nonmyeloablative Peripheral Blood Mobilized Hematopoietic Precursor Cell Transplantation for Sickle Cell Disease and Beta-Thalassemia in Individuals With Higher Risk of Transplant Failure
Brief Title: Nonmyeloablative Peripheral Blood Mobilized Hematopoietic Precursor Cell Transplantation for Sickle Cell Disease and Beta-thalassemia in People With Higher Risk of Transplant Failure
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 140077; 14-H-0077
Record Dates: First submitted 2014-04-01; First posted 2014-04-07 (Estimated); Results first posted 2024-11-29 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Sickle Cell Disease; Thalassemia; Stem Cell Transplantation; Graft vs Host Disease
Keywords: Sickle Cell Disease; Allogeneic Hematopoietic Stem Cell Transplant; Pentostatin (Nipent); Cyclophosphamide; Alemtuzumab (Campath)
MeSH Terms: conditions — Anemia, Sickle Cell; Thalassemia; Graft vs Host Disease | interventions — Alemtuzumab; Sirolimus; Cyclophosphamide; Pentostatin; Radiotherapy; Filgrastim

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Female participants with SCD or Beta-thalassemia receiving stem cell transplant with male donor (Experimental): Female participants with Sickle Cell Disease (SCD) or Beta-thalassemia receiving stem cell transplant with male donor. Pentostatin given on days -21, -17, -13, -9 and oral cyclophosphamide from days -21 to -8, with the intention to be administered in the outpatient setting. Alemtuzumab on days 7 to 3, and 300 cGy TBI on day 2. Sirolimus started at a loading dose of 5mg PO every 4 hours for three doses on day -1 and adjusted to maintain trough levels between 10-15 ng/mL. The PBSC graft targeted to deliver .10 x 106 CD34+ cells/kg (minimum .5 x 106) and infused on day 0.
  Interventions: Drug: Alemtuzumab; Drug: Sirolimus; Drug: Cyclophosphamide; Drug: Pentostatin; Procedure: Radiotherapy
- Participants with pre-existing antibodies and SCD or Beta-thalassemia receiving stem cell transplant (Experimental): Participants with pre-existing antibodies and Sickle Cell Disease (SCD) or Beta-thalassemia receiving stem cell transplant. Pentostatin given on days -21, -17, -13, -9 and oral cyclophosphamide from days -21 to -8, with the intention to be administered in the outpatient setting. Alemtuzumab on days 7 to 3, and 300 cGy TBI on day 2. Sirolimus started at a loading dose of 5mg PO every 4 hours for three doses on day -1 and adjusted to maintain trough levels between 10-15 ng/mL. The PBSC graft targeted to deliver .10 x 106 CD34+ cells/kg (minimum .5 x 106) and infused on day 0.
  Interventions: Drug: Alemtuzumab; Drug: Sirolimus; Drug: Cyclophosphamide; Drug: Pentostatin; Procedure: Radiotherapy
- Human Leukocyte Antigens (HLA) Matched Related Stem Cell Donor (Other): Participants received filgrastim to mobilize peripheral blood stem cells for apheresis collection. Collected stem cells of donor will then be infused to HLA matched sibling.
  Interventions: Drug: Filgrastim

INTERVENTIONS:
Drug: Alemtuzumab — Immunosuppressant
  Other Names: Campath
  Arms: Female participants with SCD or Beta-thalassemia receiving stem cell transplant with male donor; Participants with pre-existing antibodies and SCD or Beta-thalassemia receiving stem cell transplant
Drug: Sirolimus — Immunosuppressant
  Other Names: Rapamune
  Arms: Female participants with SCD or Beta-thalassemia receiving stem cell transplant with male donor; Participants with pre-existing antibodies and SCD or Beta-thalassemia receiving stem cell transplant
Drug: Cyclophosphamide — Immunosuppressant
  Other Names: Cytoxan
  Arms: Female participants with SCD or Beta-thalassemia receiving stem cell transplant with male donor; Participants with pre-existing antibodies and SCD or Beta-thalassemia receiving stem cell transplant
Drug: Pentostatin — Immunosuppressant
  Other Names: Deoxycoformycin
  Arms: Female participants with SCD or Beta-thalassemia receiving stem cell transplant with male donor; Participants with pre-existing antibodies and SCD or Beta-thalassemia receiving stem cell transplant
Procedure: Radiotherapy — Immunosuppressant and myelosuppressant
  Arms: Female participants with SCD or Beta-thalassemia receiving stem cell transplant with male donor; Participants with pre-existing antibodies and SCD or Beta-thalassemia receiving stem cell transplant
Drug: Filgrastim — mobilize peripheral blood stem cells for apheresis collection
  Other Names: Neupogen
  Arms: Human Leukocyte Antigens (HLA) Matched Related Stem Cell Donor

SUMMARY:
Background:

- Some sickle cell disease or beta-thalassemia can be cured with transplant. Researchers want to test a variation of transplant that uses low dose radiation and a combination of immunosuppressive drugs. They want to know if it helps a body to better accept donor stem cells.

Objectives:

- To see if low dose radiation (300 rads), oral cyclophosphamide, pentostatin, and sirolimus help a body to better accept donor stem cells.

Eligibility:

- People 4 and older with beta-thalassemia or sickle cell disease that can be cured with transplant, and their donors.

Design:

* Participants and donors will be screened with medical history, physical exam, blood test, tissue and blood typing, and bone marrow sampling. They will visit a social worker.
* Donors:
* may receive an intravenous (IV) tube in their groin vein.
* will receive a drug injection daily for 5 or 6 days to move the blood stem cells from the bone marrow into general blood circulation.
* will undergo apheresis: an IV is put into a vein in each arm. Blood is taken from one arm, a machine removes the white blood cells that contain blood stem cells, and the rest is returned through the other arm.
* Participants:
* may undergo red cell exchange procedure.
* will remain in the hospital for about 30 days.
* will receive a large IV line that can stay in their body from transplant through recovery.
* will receive a dose of radiation, and transplant related drugs by mouth or IV.
* will receive blood stem cells over 8 hours by IV.
* will take neuropsychological tests and may complete questionnaires throughout the transplant process.
* must stay near NIH for 4 months. They will visit the outpatient clinic weekly.

DETAILED DESCRIPTION:
Our ongoing nonmyeloablative allogeneic peripheral blood stem cell (PBSC) transplant protocol (03-H-0170) for patients with severe sickle cell disease (SCD) and B-thalassemia from HLA-matched family donors has excellent results thus far. Our long term leukocyte engraftment rate is 85-90% with the same disease-free survival. None of the engrafted patients had acute sickle-related events, significant toxicity associated with the conditioning regimen, or any evidence of graft versus host disease (GVHD).

While these results rival the transplant outcomes from low risk transplant patients with B-thalassemia, there are areas for improvement. The first is the 10-15% graft rejection rate, where a majority of these individuals were male donor and female recipient pairs. Another limitation is the significant delay in donor red cell engraftment in one recipient who had pre-existing allo-antibody to donor red cells from previous transfusions. Also we have excluded another group of individuals with preformed antibodies, recipients having major ABO incompatibility to the donors.

To overcome these limitations (and reduce the transplant failure rate) in this new protocol, we will continue our nonmyeloablative approach in the patients with SCD and B-thalassemia with HLA-matched family donors, but using an increased intensity regimen in a subset considered at high risk for transplant failure. This modified regimen consists of pentostatin and oral cyclophosphamide, which we hypothesize will reduce both the T cells that mediate leukocyte rejection and the B/plasma cells that produce anti-donor erythrocyte antibodies. The main transplant backbone will remain as alemtuzumab, low dose total body irradiation of 300 cGy, and sirolimus; the transplant graft will remain as unmanipulated G-CSF mobilized, T-cell replete, PBSC product for hematopoietic and lymphoid reconstitution.

The primary endpoint of this study is the percentage/number of patients who have sustained donor type hemoglobin at 1 year post transplant for male donors - female recipients. The primary endpoint for those with pre-existing antibodies is the presence of donor red cells with reticulocytes greater than or equal to 30 k/uL at 2 years post-transplant. Other endpoints include the toxicity of the pentostatin-cyclophosphamide regimen, the degree of donor-host chimerism necessary for long-term graft survival and disease amelioration, incidence of acute and chronic GVHD, incidence of graft rejection, transplant-related morbidity, as well as disease-free and overall survival. Since SCD and B-thalassemia are non-malignant disorders of red cells, severe GVHD, lack of donor erythrocyte (prolonged donor red cell aplasia), or graft rejection is collectively considered transplant failure.

ELIGIBILITY:
-INCLUSION CRITERIA- recipients (must fulfill one disease category in 1 and all of 2)

1. Disease specific

   Patients with severe sickle cell disease (not limited to Hb SS, SC, or S beta-thal) at high risk for disease-related morbidity or mortality, defined by having severe end-organ damage (A, B, C, D, or E) or potentially modifiable complication(s) not ameliorated by hydroxyurea or sickle specific therapy (F):

   --A. Stroke defined as a clinically significant neurologic event that is accompanied by an infarct on cerebral MRI or cerebral arteriopathy requiring chronic transfusion therapy; OR

   --B. Sickle cell-related renal insufficiency defined by a creatinine level greater than or equal to 1.5 times the upper limit of normal and kidney biopsy consistent with sickle cell nephropathy OR nephrotic syndrome OR creatinine clearance less than < 50mL/min OR requiring peritoneal or hemodialysis; OR

   --C. Tricuspid regurgitant jet velocity (TRV) of greater than or equal to 2.5 m/s 40, 41 at baseline; OR

   --D. Recurrent priapism defined as at least 2 episodes of an erection lasting >4 hours involving the corpora cavernosa and corpus spongiosa; OR

   --E. Sickle hepatopathy defined as EITHER ferritin >1000mcg/L OR direct bilirubin >0.4 mg/dL at baseline

   --F. Any one of the below complications:

   ---Complication/ Eligible for hydroxyurea*/ Eligible for HSCT

   ----Vaso-occlusive crises/ At least 3 hospital admissions in the last year/ More than one hospital admission in the last year while on therapeutic dose of hydroxyurea or sickle cell therapy
   * Acute chest syndrome/ 2 prior ACS/ any ACS while on hydroxyurea
   * Osetonecrosis of 2 or more joints/ And significantly affecting their quality of life by Karnofsky score 50-60/ And on hydroxyurea where total hemoglobuin increases less than 1 g/dL or fetal hemoglobin increases less than 2.5 times the baseline level
   * Red cell alloimmunization/ Transfusion dependent/ Total hemoglobin increases less than 1g/dL while on hydroxurea

     2. Patients with beta-thalassemia who have grade 2 or 3 iron overload, determined by the presence of 2 or more of the following:

     -- portal fibrosis by liver biopsy
     * inadequate chelation history (defined as failure to maintain adequate compliance with chelation with deferoxamine initiated within 18 months of the first transfusion and administered subcutaneously for 8-10 hours at least 5 days each week)
     * hepatomegaly of greater than 2cm below the costochondral margin

   Non-disease specific:

   -Age greater than or equal to 4 years

   -6/6 HLA matched family donor available
   * Ability to comprehend and willing to sign an informed consent
   * Negative beta-HCG, when applicable

   EXCLUSION CRITERIA -recipient (any of the following would exclude the subject from participating)

   -ECOG performance status of 3 or more

   -Evidence of uncontrolled bacterial, viral, or fungal infections (currently taking medication and progression of clinical symptoms) within one month prior to starting the conditioning regimen. Patients with fever or suspected minor infection should await resolution of symptoms before starting the conditioning regimen.

   -Major anticipated illness or organ failure incompatible with survival from PBSC transplant

   -Pregnant or lactating

   INCLUSION CRITERIA -donor

   -6/6 HLA matched family donor deemed suitable and eligible, and willing to donate, per clinical evaluations who are additionally willing to donate blood for research. Matched related donors will be evaluated in accordance with existing Standard NIH Policies and Procedures for determination of eligibility and suitability for clinical donation. Note that participation in this study is offered to all matched related donors, but is not required for a donor to make a stem cell donation, so it is possible that not all related donors will enroll onto this study.

   EXCLUSION CRITERIA -donor

   -None

Ages: 4 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2014-04-21 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2027-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew M Hsieh, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF
Time Frame: At the time of publication or by the end of the protocol, whichever comes first, and available indefinitely
Access Criteria: Data will be shared upon request by sending a request to matthewhs@nhlbi.nih.gov

REFERENCES:
- [Derived] Inam Z, Jeffries N, Link M, Coles W, Pollack P, Luckett C, Phang O, Harvey E, Martin T, Farrey T, Tisdale JF, Hsieh MM. Two Nonmyeloablative HLA-Matched Related Donor Allogeneic Hematopoietic Cell Transplantation Regimens in Patients with Severe Sickle Cell Disease. Transplant Cell Ther. 2025 May;31(5):305-318. doi: 10.1016/j.jtct.2025.02.021. Epub 2025 Feb 24. PMID 40010689
- [Derived] Leonard A, Furstenau D, Abraham A, Darbari DS, Nickel RS, Limerick E, Fitzhugh C, Hsieh M, Tisdale JF. Reduction in vaso-occlusive events following stem cell transplantation in patients with sickle cell disease. Blood Adv. 2023 Jan 24;7(2):227-234. doi: 10.1182/bloodadvances.2022008137. PMID 36240296
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2014-H-0077.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Female Participants With SCD or Beta-thalassemia Receiving Stem Cell Transplant With Male Donor | Participants With Pre-existing Antibodies and SCD or Beta-thalassemia Receiving Stem Cell Transplant | Human Leukocyte Antigens (HLA) Matched Related Stem Cell Donor
Started | 11 | 18 | 27
Completed | 7 | 16 | 27
Not Completed | 4 | 2 | 0
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Death | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Female Participants With SCD or Beta-thalassemia Receiving Stem Cell Transplant With Male Donor | Participants With Pre-existing Antibodies and SCD or Beta-thalassemia Receiving Stem Cell Transplant | Human Leukocyte Antigens (HLA) Matched Related Stem Cell Donor | Total
Number analyzed (Participants) | 11 | 18 | 27 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 3 | 5 | 8
  Between 18 and 65 years | 11 | 15 | 22 | 48
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 8 | 24
  Male | 0 | 13 | 19 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 17 | 25 | 52
  Unknown or Not Reported | 1 | 1 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 16 | 23 | 49
  White | 0 | 0 | 0 | 0
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 11 | 18 | 27 | 56

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Have Sustained Donor Type Hemoglobin at One Year Post Transplant
Description: Number of patients who have sustained donor type hemoglobin at one year post transplant. Sustained donor type hemoglobin is based on hemoglobin electrophoresis for patients with SCD and transfusion independence for patients with beta-thalassemia
Time Frame: 1 year
Population: Analysis is intended per protocol for cohort 1 participants that received a stem cell transplant (female participants with male donors)
Measure: Count of Participants; unit: Participants
Arm/Group | Female Participants With SCD or Beta-thalassemia Receiving Stem Cell Transplant With Male Donor
Number analyzed (Participants) | 11
Participants | 10

2. Primary Outcome: Number of Participants With Donor Red Cells at 2 Years Post Stem Cell Transplant
Description: Number of participants with donor red cells at 2 years post stem cell transplant. Number of participants with donor red cells is detected by hemoglobin electrophoresis or donor type red cell antigen, and reticulocyte count ≥30 k/uL at 2 years post-transplant.
Time Frame: 2 years
Population: Analysis is intended per protocol to include those participants from cohort 2 (patients with pre-existing antibody to donor red cells)
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Pre-existing Antibodies and SCD or Beta-thalassemia Receiving Stem Cell Transplant
Number analyzed (Participants) | 18
Participants | 16

3. Secondary Outcome: Mean CD34+ Cell Dose
Description: Mean CD34+ cell dose, filgrastim mobilized peripheral blood hematopoietic cells, unselected
Time Frame: Day 0 up to Day 1
Measure: Mean (Standard Deviation); unit: x10^6 cells/kg
Arm/Group | Female Participants With SCD or Beta-thalassemia Receiving Stem Cell Transplant With Male Donor | Participants With Pre-existing Antibodies and SCD or Beta-thalassemia Receiving Stem Cell Transplant
Number analyzed (Participants) | 11 | 18
x10^6 cells/kg | 19.08 (8.38) | 14.98 (5.95)

4. Secondary Outcome: Mean CD3+ Cell Dose
Description: Mean CD3+ cell dose, filgrastim mobilized peripheral blood hematopoietic cells, unselected
Time Frame: Day 0 up to Day 1
Measure: Mean (Standard Deviation); unit: x10^8 cells/kg
Arm/Group | Female Participants With SCD or Beta-thalassemia Receiving Stem Cell Transplant With Male Donor | Participants With Pre-existing Antibodies and SCD or Beta-thalassemia Receiving Stem Cell Transplant
Number analyzed (Participants) | 11 | 18
x10^8 cells/kg | 3.12 (1.37) | 3.29 (1.57)

5. Secondary Outcome: Median Percent of Donor T-cells and Myeloid Chimerism
Description: Median Percent of donor T-cells and myeloid chimerism. Leukocytes are selected by magnetic beads for CD3 (T-cells) and CD14/15 (myeloid cells), then microsatellite PCR analyses are performed to obtain donor chimerism percent.
Time Frame: day 30, day 60 , day 100, 1 year and 2 year
Population: Analysis includes those participants who have sustained engraftment or did not experience graft failure.
Measure: Median (Full Range); unit: percentage of donor cells
Arm/Group | Female Participants With SCD or Beta-thalassemia Receiving Stem Cell Transplant With Male Donor | Participants With Pre-existing Antibodies and SCD or Beta-thalassemia Receiving Stem Cell Transplant
Number analyzed (Participants) | 10 | 16
percentage of donor cells
  myeloid chimerism D30 | 100 [80 to 100] | 99.5 [68 to 100]
  myeloid chimerism D60 | 100 [54 to 100] | 100 [29 to 100]
  myeloid chimerism D100 | 100 [42 to 100] | 100 [16 to 100]
  myeloid chimerism Year 1 | 100 [47 to 100] | 100 [54 to 100]
  myeloid chimerism Year 2 | 100 [44 to 100] | 99 [45 to 100]
  donor T-cells D30 | 65.5 [16 to 94] | 25 [1 to 85]
  donor T-cells D60 | 39 [2 to 86] | 23 [1 to 100]
  donor T-cells D100 | 34 [0 to 91] | 22.5 [2 to 96]
  donor T-cells Year 1 | 70 [29 to 78] | 43 [24 to 100]
  donor T-cells Year 2 | 74.5 [53 to 84] | 62 [27 to 94]

6. Secondary Outcome: Number of Participants Who Developed Acute Graft vs Host Disease (GVHD) Grades I, II, III, IV
Description: Number of participants who developed Acute Graft vs Host Disease (GVHD) Grades I, II, III, IV as defined by CIMBTR criteria for Organ Stages of Acute GVHD.
  Grades are defined as:
  Grade I: Skin = Maculopapular rash< 25% of body surface area (BSA); Liver = Total Bilirubin 2-3 mg/dL; Lower GI = stool output/day is 500-999 mL/day.
  Grade II: Skin = rash on 25-50 percent body surface area; Liver = Total Bilirubin 3.1-6.0 mg/dL; Lower GI = Diarrhea 1001-1500 mL/day.
  Grade III: Skin = Rash on >50% of body surface; Liver = Total Bilirubin 6.1 - 15.0 mg/dL; Lower GI = Diarrhea > 1500 mL/day.
  Grade IV: Skin = Generalized erythroderma plus bullous formation; Liver = Total Bilirubin >15 mg/dL; Lower GI = Severe abdominal pain with or without ileus.
  Grade I GVHD is characterized as mild disease, grade II GVHD as moderate, grade III as severe, and grade IV life-threatening.
Time Frame: Up to Day 100
Population: Analysis includes those participants who have sustained engraftment or did not experience graft failure.
Measure: Count of Participants; unit: Participants
Arm/Group | Female Participants With SCD or Beta-thalassemia Receiving Stem Cell Transplant With Male Donor | Participants With Pre-existing Antibodies and SCD or Beta-thalassemia Receiving Stem Cell Transplant
Number analyzed (Participants) | 10 | 16
Participants
  Grade I | 0 | 0
  Grade II | 0 | 1
  Grade III | 1 | 0
  Grade IV | 0 | 0

7. Secondary Outcome: Number of Participants Who Developed Moderate or Severe Chronic Graft vs Host Disease (GVHD)
Description: Number of Participants Who Developed Moderate or Severe Chronic Graft vs Host Disease (GVHD) up to 5 years.
  Moderate chronic GVHD involves EITHER 3 organs/sites with no clinically significant functional impairment OR a less than or equal to 1 organ/site with clinically significant functional impairment, but no major disability. Severe GVHD is associated with a major disability caused by chronic GVHD.
Time Frame: Day 100 up to 2 years
Population: Analysis includes those participants who have sustained engraftment or did not experience graft failure.
Measure: Count of Participants; unit: Participants
Arm/Group | Female Participants With SCD or Beta-thalassemia Receiving Stem Cell Transplant With Male Donor | Participants With Pre-existing Antibodies and SCD or Beta-thalassemia Receiving Stem Cell Transplant
Number analyzed (Participants) | 10 | 16
Participants
  Moderate | 0 | 0
  Severe | 0 | 0

8. Secondary Outcome: Number of Participants That Experienced Graft Failure or Graft Rejection, or Red Cell Aplasia at 2 Years After Transplant
Description: Number of participants that experienced graft failure or graft rejection, or red cell aplasia at 2 years after transplant. Graft failure or graft rejection is defined as <5% donor cells in both CD3 and myeloid chimerism. Red cell aplasia is defined as reticulocyte <30 k/uL and requiring red cell transfusions.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Female Participants With SCD or Beta-thalassemia Receiving Stem Cell Transplant With Male Donor | Participants With Pre-existing Antibodies and SCD or Beta-thalassemia Receiving Stem Cell Transplant
Number analyzed (Participants) | 11 | 18
Participants
  graft failure | 1 | 0
  red cell aplasia | 0 | 2

9. Secondary Outcome: Number of Participants That Experienced Regimen Failure
Description: Number of Participants That Experienced Regimen Failure. Regimen failure is defined as those participants that experienced grade 3 or higher acute GVHD, moderate/severe chronic GVHD, graft failure/rejection, or red cell aplasia. Together any one of these count toward the combined endpoint of regimen failure.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Female Participants With SCD or Beta-thalassemia Receiving Stem Cell Transplant With Male Donor | Participants With Pre-existing Antibodies and SCD or Beta-thalassemia Receiving Stem Cell Transplant
Number analyzed (Participants) | 11 | 18
Participants | 2 | 2

10. Secondary Outcome: Number of Participants That Experienced Transplant-related Mortality
Description: Number of participants that experienced transplant-related mortality. Transplant-related mortality is defined as death that is at least possibly related to the transplant (GVHD, toxicity, infection, other causes).
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Female Participants With SCD or Beta-thalassemia Receiving Stem Cell Transplant With Male Donor | Participants With Pre-existing Antibodies and SCD or Beta-thalassemia Receiving Stem Cell Transplant
Number analyzed (Participants) | 11 | 18
Participants | 0 | 0

11. Secondary Outcome: Percentage of Participant With Disease-free Survival Following Stem Cell Transplant
Description: Percentage of participant with disease-free survival following stem cell transplant. Disease-free survival is defined as alive and free acute complications related to sickle cell disease.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Female Participants With SCD or Beta-thalassemia Receiving Stem Cell Transplant With Male Donor | Participants With Pre-existing Antibodies and SCD or Beta-thalassemia Receiving Stem Cell Transplant
Number analyzed (Participants) | 11 | 18
Participants | 9 | 16

12. Secondary Outcome: Percentage of Participant Overall Survival Following Stem Cell Transplant
Description: Percentage of Participant Overall Survival up to year 2 following stem cell transplant. Overall survival is defined as being alive following stem cell transplant.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Female Participants With SCD or Beta-thalassemia Receiving Stem Cell Transplant With Male Donor | Participants With Pre-existing Antibodies and SCD or Beta-thalassemia Receiving Stem Cell Transplant
Number analyzed (Participants) | 11 | 18
Participants | 10 | 17

13. Secondary Outcome: Median Day to Neutrophil Recovery
Description: Median Day to Neutrophil recovery. Neutrophil recovery is defined as the first of three consecutive days of neutrophil count >0.5 x 10^9 cells/uL.
Time Frame: Up to Day 100
Measure: Median (Full Range); unit: days
Arm/Group | Female Participants With SCD or Beta-thalassemia Receiving Stem Cell Transplant With Male Donor | Participants With Pre-existing Antibodies and SCD or Beta-thalassemia Receiving Stem Cell Transplant
Number analyzed (Participants) | 11 | 18
days | 22 [17 to 67] | 20.5 [8 to 25]

14. Secondary Outcome: Median Days to Platelet Recovery
Description: Median Days to Platelet Recovery. Platelet recovery is defined as count >50 cells/uL and 7 days from the last platelet transfusion.
Time Frame: Up to Day 120
Measure: Median (Full Range); unit: days
Arm/Group | Female Participants With SCD or Beta-thalassemia Receiving Stem Cell Transplant With Male Donor | Participants With Pre-existing Antibodies and SCD or Beta-thalassemia Receiving Stem Cell Transplant
Number analyzed (Participants) | 11 | 18
days | 21.5 [16 to 69] | 22.5 [10 to 112]

15. Secondary Outcome: Median Days to Red Cell Recovery
Description: Median Days to Red Cell Recovery. Red cell recovery defined as days to recovery of reticulocyte count .30 k/uL, detection of donor red cells, transfusion independence.
Time Frame: Up to 2 years
Measure: Median (Full Range); unit: days
Arm/Group | Female Participants With SCD or Beta-thalassemia Receiving Stem Cell Transplant With Male Donor | Participants With Pre-existing Antibodies and SCD or Beta-thalassemia Receiving Stem Cell Transplant
Number analyzed (Participants) | 11 | 18
days | 22 [15 to 75] | 19 [8 to 195]

ADVERSE EVENTS:
Time Frame: 5 years
Description: Information on AEs will be solicited from subjects through questions from study personnel and/or information volunteered by the subject. Grade 3 or higher adverse event recording will start at the time of conditioning regimen, will be followed until satisfactory resolution, through final study visit.
Arm/Group | Female Participants With SCD or Beta-thalassemia Receiving Stem Cell Transplant With Male Donor | Participants With Pre-existing Antibodies and SCD or Beta-thalassemia Receiving Stem Cell Transplant | Human Leukocyte Antigens (HLA) Matched Related Stem Cell Donor
All-Cause Mortality (participants affected / at risk) | 1/11 | 1/18 | 0/27
Serious Adverse Events (participants affected / at risk) | 9/11 | 13/18 | 2/27
Other Adverse Events (participants affected / at risk) | 11/11 | 18/18 | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Female Participants With SCD or Beta-thalassemia Receiving Stem Cell Transplant With Male Donor (N=11) | Participants With Pre-existing Antibodies and SCD or Beta-thalassemia Receiving Stem Cell Transplant (N=18) | Human Leukocyte Antigens (HLA) Matched Related Stem Cell Donor (N=27)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 2 (5) | 0 (0) | 0 (0)
Bacteremia (Infections and infestations) | 3 (6) | 0 (0) | 0 (0)
Clostridioides difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Cytomegalovirus (CMV) Reactivation (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epstein-Barr virus (EBV) viremia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Micro Papillary Thyroid Carcinoma (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 2 (2) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Herpes simplex reactivation (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (4) | 0 (0)
Hypokalemia (Investigations) | 1 (7) | 0 (0) | 0 (0)
Typhoid fever (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Malaria (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Lung infection (Infections and infestations) | 3 (3) | 1 (2) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (Musculoskeletal and connective tissue disorders) | 2 (11) | 6 (8) | 1 (1)
Vaso-occlusive pain crisis (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (5) | 0 (0)
Psychosis (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Furunculosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Liver biopsy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Plasma exchange (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Teeth extractions (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Hip replacement (Surgical and medical procedures) | 0 (0) | 1 (2) | 0 (0)
Tunneled catheter removal (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Tunneled line insertion (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Wound care (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
White blood cell decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Headache (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Emesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypocalcemia (Investigations) | 0 (0) | 0 (0) | 2 (2)
Hypomagnesemia (Investigations) | 0 (0) | 0 (0) | 2 (2)
Hypophosphatemia (Investigations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Female Participants With SCD or Beta-thalassemia Receiving Stem Cell Transplant With Male Donor (N=11) | Participants With Pre-existing Antibodies and SCD or Beta-thalassemia Receiving Stem Cell Transplant (N=18) | Human Leukocyte Antigens (HLA) Matched Related Stem Cell Donor (N=27)
Acute GVHD (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 5 (8) | 0 (0)
CD4 lymphocytes decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 3 (5) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 9 (16) | 10 (25) | 0 (0)
Neutrophil count decreased (Blood and lymphatic system disorders) | 8 (15) | 8 (28) | 0 (0)
Platelet count decreased (Blood and lymphatic system disorders) | 6 (9) | 5 (11) | 0 (0)
White blood cell decreased (Blood and lymphatic system disorders) | 5 (6) | 2 (4) | 0 (0)
Hypertension (Cardiac disorders) | 2 (2) | 4 (4) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Hemianopsia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (2) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Agitation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1) | 0 (0)
Infusion related reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 2 (7) | 0 (0) | 0 (0)
Pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 6 (13) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypogammaglobulinemia (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Anorectal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Cytomegalovirus (CMV) Reactivation (Infections and infestations) | 3 (3) | 4 (6) | 0 (0)
Endocarditis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
BK Virus Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Methicillin-resistant Staphylococcus aureus (MRSA) infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasal vestibulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (3) | 0 (0)
Hyperuricemia (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Investigations) | 0 (0) | 1 (2) | 0 (0)
Hypophosphatemia (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Iron overload (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0)
Obsessive-compulsive disorder (OCD) (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Pseudoseizure (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Right Heart Catheterization (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Thyroidectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphedema (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-13): https://cdn.clinicaltrials.gov/large-docs/66/NCT02105766/Prot_SAP_000.pdf